CLINICAL TRIAL: NCT04235608
Title: Sevoflurane for Sedation in Acute Respiratory Distress Syndrome: a Multicenter Prospective Randomized Trial
Brief Title: SEvoflurane for Sedation in ARds
Acronym: SESAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SESAR - RBHP 2018 JABAUDON
Record Dates: First submitted 2020-01-14; First posted 2020-01-22 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-06

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: ARDS; Sedation; Inhaled sevoflurane
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Intervention Model Description: Investigator-initiated, multicenter, prospective, randomized, stratified, parallel-group clinical trial with blinded outcome assessment and concealed allocation of patients with moderate-to-severe ARDS to a strategy of inhaled sedation with sevoflurane or to a strategy of current intravenous sedation practice using propofol.
Who Masked: Outcomes Assessor
Masking Description: At each participating center, patients will be followed up for primary and secondary endpoints by members of the research staff who will be unaware of the trial group allocation. Information on whether the primary and secondary outcomes occur will be collected and entered into the electronic web-based case report form (eCRF) by trial or clinical trained personal (clinical research associate), blinded to the allocation group, under the supervision of the local principal investigator (PI) or designee who will also be unaware of the trial group allocation.
  Finally, the independent trial statistician and the members of the data monitoring and safety committee (DMSC) will also remain blinded for the allocation during analysis. However, the observation of differences in serious adverse events between the two groups will allow, for safety reasons may the DMSC deem necessary, to unblind allocation groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- inhaled sedation with sevoflurane (Experimental): Inhaled sedation with sevoflurane, as vaporized via the Anesthesia Conserving Device (AnaConDa-S, Sedana Medical, Danderyd, Sweden)
  Interventions: Drug: Inhaled sedation with sevoflurane
- intravenous sedation with propofol (Active Comparator): intravenous sedation with propofol, as already routinely used in participating ICUs
  Interventions: Drug: intravenous sedation with propofol

INTERVENTIONS:
Drug: Inhaled sedation with sevoflurane — Inhaled sedation with sevoflurane using the Anesthesia Conserving Device (AnaConDa-S, Sedana Medical, Danderyd, Sweden).
  Arms: inhaled sedation with sevoflurane
Drug: intravenous sedation with propofol — intravenous sedation with propofol, as already routinely used in participating ICUs.
  Arms: intravenous sedation with propofol

SUMMARY:
This study evaluates whether a sedation with inhaled sevoflurane will decrease mortality and increase time off the ventilator at 28 days in patients with acute respiratory distress syndrome (ARDS).

Half of the patients will receive inhaled sedation with sevoflurane and the other half will receive intravenous sedation with propofol.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

To assess the efficacy of a sedation with inhaled sevoflurane in improving in reducing mortality and morbidity in patients with moderate-severe ARDS in comparison to a control group receiving intravenous sedation with propofol.

PRIMARY HYPOTHESIS:

Inhaled sedation with sevoflurane will improve a composite outcome of mortality and time off the ventilator at 28 days, in patients with moderate-severe ARDS.

The trial will accrue a maximum of 700 patients. Patients will be recruited from participating intensive care units and randomized to the active (inhaled sevoflurane) or control (intravenous propofol).

The overall strategy is to screen and enroll early, every newly intubated, acutely ill or postoperative, patient at each site, using clinically obtained pulse oximetry and blood gases.

By providing superior awakening and extubation times, as well as lung-protective effects from anti-inflammatory and protective effects from epithelial injury, inhaled sevoflurane may hasten recovery from lung injury and improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Presence for ≤24 hours of all of the following conditions, within one week of a clinical insult or new or worsening respiratory symptoms:

  * PaO2/FiO2 <150 mmHg with positive end-expiratory pressure (PEEP) ≥8 cmH2O (or, if arterial blood gas not available, SpO2/FiO2 that is equivalent to a PaO2/FiO2 <150 mmHg with PEEP ≥8 cmH2O and a confirmatory SpO2/FiO2 between 1-6 hours after the initial SpO2/FiO2 determination)
  * Bilateral opacities not fully explained by effusions, lobar/lung collapse, or nodules
  * Respiratory failure not fully explained by cardiac failure or fluid overload; need objective assessment (e.g., echocardiography) to exclude hydrostatic edema if no risk factor present

Exclusion Criteria:

* Absence of affiliation to the French Sociale security
* Patient under a tutelage measure or placed under judicial protection
* Continuous sedation with inhaled sevoflurane at enrollment
* Known pregnancy
* Currently receiving ECMO therapy
* Chronic respiratory failure defined as PaCO2 >60 mmHg in the outpatient setting
* Home mechanical ventilation (non-invasive ventilation or via tracheotomy) except for CPAP/BIPAP used solely for sleep-disordered breathing
* Body mass index >40 kg/m2
* Chronic liver disease defined as a Child-Pugh score of 12-15
* Expected duration of mechanical ventilation <48 hours
* Moribund patient, i.e. not expected to survive 24 hours despite intensive care
* Burns >70% total body surface
* Previous hypersensitivity or anaphylactic reaction to sevoflurane or cisatracurium
* Medical history of malignant hyperthermia
* Long QT syndrome at risk of arrhythmic events
* Medical history of liver disease attributed to previous exposure to a halogenated agent (including sevoflurane)
* Known hypersensitivity to propofol or any of its components
* Known allergy to eggs, egg products, soybeans, and soy products
* Suspected or proven intracranial hypertension
* Tidal volume of 6 mL/kg predicted body weight (PBW) below 200 mL (as recommended by the manufacturer for the use of the AnaConDa-S (Sedana Medical, Danderyd, Sweden)
* Enrollment in another interventional ARDS trial with direct impact on sedation and mechanical ventilation
* Endotracheal ventilation for greater than 120 hours (5 days)
* Persistent bronchopleural fistula despite chest tube drainage
* PaO2/FiO2 (if available) >200 mmHg after meeting inclusion criteria and before randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2020-05-03 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
Ventilator-free days through day 28 | Day 28
  Number of days alive and off the ventilator at 28 days, thereby considering death as a competing event

SECONDARY OUTCOMES:
90-day survival (Key secondary outcome) | Day 90
All-cause, all-location 28-day mortality (Secondary outcome) | Day 28
All-cause hospital 28-day mortality (Secondary outcome) | Day 28
All-cause, all-location 14-day mortality (Secondary outcome) | Day 14
All-cause, all-location 7-day mortality (Secondary outcome) | Day 7

OTHER OUTCOMES:
Ventilator-free days through day 14 (Exploratory outcome) | Day 14
  Number of days alive and off the ventilator at 14 days, thereby considering death as a competing event
Ventilator-free days through day 7 (Exploratory outcome) | Day 7
  Number of days alive and off the ventilator at 7 days, thereby considering death as a competing event
Organ failure-free days through day 7 (Exploratory outcome) | Day 7
  Organ failure is defined as present on any date when the most abnormal vital signs or clinically available lab value meets the definition of clinically significant organ failure according to SOFA scores. Patients will be followed for development of organ failures to death, hospital discharge or study day 7, whichever comes first. Each day a patient is alive and free of a given organ failure will be scored as a failure-free day. Any day that a patient is alive and free of all organ failures will represent days alive and free of all organ failure.
ICU-free days through day 28 (Exploratory outcome) | Day 28
Hospital-free days through day 28 (Exploratory outcome) | Day 28
Changes in oxygenation index through day 7 (Exploratory outcome) | Day 7
Changes in PaO2/FiO2 through day 7 (Exploratory outcome) | Day 7
Changes in PaCO2 through day 7 (Exploratory outcome) | Day 7
Changes in arterial pH through day 7 (Exploratory outcome) | Day 7
Changes in PEEP through day 7 (Exploratory outcome) | Day 7
Changes in inspiratory plateau pressure through day 7 (Exploratory outcome) | Day 7
Changes in static compliance of the respiratory system through day 7 (Exploratory outcome) | Day 7
Changes in ventilatory ratio through day 7 (Exploratory outcome) | Day 7
Use of rescue procedures for refractory hypoxemia through day 28 (Exploratory outcome) | Day 28
  Rescue procedures will be chosen according to the practice at clinical sites: nitric oxide, epoprostenol sodium, high frequency ventilation, use of neuromuscular blockade after 48 h from randomization, and extracorporeal membrane oxygenation.
ICU-acquired delirium through day 7 (Exploratory outcome) | Day 7
  Confusion Assessment Method for the ICU (CAM-ICU) assessed daily from study entry to study day 7, death or ICU discharge, whichever comes first.
Disability at 3 months (Exploratory outcome) | Day 90
  Katz Activities of Daily Living (ADL)
Disability at 12 months (Exploratory outcome) | Day 365
  Katz Activities of Daily Living (ADL)
Health-Related Quality of Life at 3 months (Exploratory outcome) | Day 90
  Short Form-36 (SF-36)
Health-Related Quality of Life at 12 months (Exploratory outcome) | Day 365
  Short Form-36 (SF-36)
Self-rated health at 3 months (Exploratory outcome) | Day 90
  Health questionnaire (1 standard item)
Self-rated health at 12 months (Exploratory outcome) | Day 365
  Health questionnaire (1 standard item)
Pain-interference at 3 months (Exploratory outcome) | Day 90
  Pain-interference (1 standard item)
Pain-interference at 12 months (Exploratory outcome) | Day 365
  Pain-interference (1 standard item)
Post-Traumatic Stress Symptoms-14 at 3 months (Exploratory outcome) | Day 90
Hospital Anxiety and Depression Scale at 3 months (Exploratory outcome) | Day 90
Post-Traumatic Stress Symptoms-14 at 12 months (Exploratory outcome) | Day 365
Hospital Anxiety and Depression Scale at 12 months (Exploratory outcome) | Day 365
Cognitive function at 3 months (Exploratory outcome) | Day 90
  Alzheimer's Disease-8
Cognitive function at 12 months (Exploratory outcome) | Day 365
  Alzheimer's Disease-8
Subsequent return to work, hospital and emergency department use, and location of residence at 3 months (Exploratory outcome) | Day 90
Subsequent return to work, hospital and emergency department use, and location of residence at 12 months (Exploratory outcome) | Day 365
Healthcare-related costs during ICU stay (Exploratory outcome) | Through study completion, an average of 1 year
Healthcare-related costs during hospital stay (Exploratory outcome) | Through study completion, an average of 1 year
Plasma biomarker levels of IL-8, sTNFr1, bicarbonates (hyperinflammatory ARDS phenotype), IL-6 (VILI), ANG-2 (endothelial activation), and sRAGE (alveolar epithelial injury) though day 14 (Exploratory biological outcome) | Day 14
  Changes over time (as measured at study entry and on days 1, 2, 4, 6 and 14 or ICU discharge, whichever occurs first)
Change in urine biomarkers of TIMP-2 and IGFBP-7 (acute kidney injury) though day 14 (Exploratory biological outcome) | Day 14
  Changes over time (as measured at study entry and on days 1, 2, 4, 6 and 14 or ICU discharge, whichever occurs first)
Change in plasma total fluoride and hexafluoroisopropanol (sevoflurane metabolism) though day 14 (Exploratory biological outcome) | Day 14
  Changes over time (as measured at study entry and on days 1, 2, 4, 6 and 14 or ICU discharge, whichever occurs first)
Genetic analysis: DNA and RNA expressions through day 2 (Exploratory biological outcome) | Day 2
  Whole blood will be collected at baseline and at 48 h for RNA and DNA studies
Total protein level within undiluted pulmonary edema fluid (alveolar fluid clearance) through day 1 (Exploratory biological outcome) | Day 1
  Undiluted pulmonary edema fluid will be collected at baseline and 24 h from 50 patients from each group
Biomarker measurements in the fluid from heat moisture exchanger filters (control group) or AnaConDa-S devices (intervention group) through day 1 (Exploratory biological outcome) | Day 1
  Heat moisture exchanger filter or AnaConDa-S devices will be collected at 24 h in 30 patients randomized to the control group and 30 patients randomized to intervention group
Biomarker measurements in the broncho-alveolar lavage fluid through day 6 (Exploratory biological outcome) | Day 6
  Broncho-alveolar lavage fluid samples will be collected from a total of 25 patients within 48 h from study entry and between day 4 and day 6 after randomization
Hemodynamic measures (mean arterial pressure) through day 7 (Safety outcome) | Day 7
Hemodynamic measures (dose of infused norepinephrine or other vasopressor) through day 7 (Safety outcome) | Day 7
Hemodynamic measures (serum lactate level) through day 7 (Safety outcome) | Day 7
Measures of renal function (KDIGO criteria for acute kidney injury) through day 7 (Safety outcome) | Day 7
Supraventricular tachycardia or new onset atrial fibrillation through day 7 (Safety outcome) | Day 7
Severe hypercapnic acidosis with arterial pH <7.15 through day 7 (Safety outcome) | Day 7
Development of malignant hyperthermia through day 7 (Safety outcome) | Day 7
Development of propofol-related infusion syndrome through day 7 (Safety outcome) | Day 7
Development of pneumothorax or bronchopleural fistula persistent despite drainage through day 7 (Safety outcome) | Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Jabaudon, Study Chair — University Hospital, Clermont-Ferrand; Raïko Blondonnet, Principal Investigator — University Hospital, Clermont-Ferrand; Jean-Michel Constantin, Principal Investigator — APHP - La Pitié Salpêtrière; Antoine Roquilly, Principal Investigator — Nantes University Hospital; Samir Jaber, Principal Investigator — CHU Montpellier - Saint-Eloi; Virginie Lemiale, Principal Investigator — APHP - Saint-Louis; Carole Ichai, Principal Investigator — CHU NICE; Lionel Velly, Principal Investigator — APHM - La Timone; Stéphanie Bulyez, Principal Investigator — CHU Nîmes; Sigismond Lasocki, Principal Investigator — University Hospital, Angers; Jean-Pierre Quenot, Principal Investigator — CHU Dijon; Thomas Lebouvier, Principal Investigator — CHU Rennes; François Legay, Principal Investigator — CH Brieuc; Arnaud W. Thille, Principal Investigator — CHU Poitiers; Alexandre Lautrette, Principal Investigator — Centre Jean-Perrin Clermont-Ferrand; Julien Pottecher, Principal Investigator — CHU Strasbourg; Franck Verdonk, Principal Investigator — APHP - Saint-Antoine; Christophe Vinsonneau, Principal Investigator — CH Béthune; Pierre-Marie Bertrand, Principal Investigator — CH Cannes; Mehran Monchi, Principal Investigator — CH Melun-Sénart; Joël Cousson, Principal Investigator — CHU REIMS; Julien Maizel, Principal Investigator — CHU Amiens; Erwan L'Her, Principal Investigator — CHU Brest; Belaïd Bouhemad, Principal Investigator — CHU Dijon; Boris Jung, Principal Investigator — CHU Montpellier - Lapeyronie; Claire Dahyot-Fizelier, Principal Investigator — CHU Poitiers; Claire Lhommet, Principal Investigator — Hopital Diaconesses - La Croix Simon; Caroline Varillon, Principal Investigator — CH Dunkerque; Arthur Durand, Principal Investigator — CHU Lille; Marc Gainnier, Principal Investigator — APHM - La Timone; Fabien Lambiotte, Principal Investigator — Hospital Valenciennes; Julien Lorber, Principal Investigator — Hospital, Saint Nazaire; Delphine Brégeaud, Principal Investigator — HOSPITAL, SAINTES; Aziz Berrouba, Principal Investigator — Hospital Martigues; Julio Badie, Principal Investigator — Hospital Belfort; Alexandre Conia, Principal Investigator — HOSPITAL, CHARTRES; François Thouy, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (33):
- France (33):
  - University Hospital, Amiens
  - University Hospital, Angers
  - Hospital Belfort, Belfort
  - Hospital, Béthune
  - Cavale Blanche Hospital - University Hospital, Brest
  - Hospital, Cannes
  - Hospital Chartres, Chartres
  - University Hospital,, Clermont-Ferrand
  - Jean Perrin Comprehensive Cancer Center, Clermont-Ferrand
  - University Hospital, Clermont-Ferrand
  - University Hospital, Dijon
  - Hospital, Dunkirk
  - Salengro Hospital - University Hospital, Lille
  - Timone Hospital - Assistance Publique-Hôpitaux, Marseille
  - Hospital Martigues, Martigues
  - Hospital, Melun
  - Lapeyronie Hospital - University Hospital, Montpellier
  - Saint-Eloi Hospital - University Hospital, Montpellier
  - Hotel Dieu Hospital - University Hospital, Nantes
  - Pasteur 2 Hospital - University Hospital, Nice
  - Carémeaux Hospital - University Hospita, Nîmes
  - Diaconesses - La Croix Simon Hospital, Paris
  - Pitié-Salpêtrière Hospital, - Assistance Publique-Hôpitaux, Paris
  - Saint-Antoine University Hospital - Assistance Publique-Hôpitaux, Paris
  - Saint-Louis University Hospital - Assistance Publique-Hôpitaux, Paris
  - University Hospital, Poitiers
  - University Hospital, Reims
  - University Hospital, Rennes
  - Hospital, Saint-Brieuc
  - Hospital Saint-Nazaire, Saint-Nazaire
  - Hospital, Saintes
  - Hautepierre Hospital, University Hospitals, Strasbourg
  - Hospital Valenciennes, Valenciennes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jabaudon M, Quenot JP, Badie J, Audard J, Jaber S, Rieu B, Varillon C, Monsel A, Thouy F, Lorber J, Cousson J, Bulyez S, Bourenne J, Sboui G, Lhommet C, Lemiale V, Bouhemad B, Brault C, Lasocki S, Legay F, Lebouvier T, Durand A, Pottecher J, Conia A, Bregeaud D, Velly L, Thille AW, Lambiotte F, L'Her E, Monchi M, Roquilly A, Berrouba A, Verdonk F, Chabanne R, Godet T, Garnier M, Blondonnet R, Vernhes J, Sapin V, Borao L, Futier E, Pereira B, Constantin JM; SESAR Trial Investigators. Inhaled Sedation in Acute Respiratory Distress Syndrome: The SESAR Randomized Clinical Trial. JAMA. 2025 May 13;333(18):1608-1617. doi: 10.1001/jama.2025.3169. PMID 40098564